CLINICAL TRIAL: NCT03750253
Title: Extracorporeal Shock Wave Therapy for Pain-Relief After Arthroscopy for Osteochondral Lesions of the Talus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Xiaojun Duan, Deputy Director of the Center for Joint Surgery, Southwest Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ESWT
Record Dates: First submitted 2018-11-18; First posted 2018-11-23 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Osteochondral Lesion of Talus
Keywords: Extracorporeal Shock Wave Therapy; Osteochondral Lesions of Talus; Arthroscopy; Pain-relief
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extracorporeal Shock Wave Therapy (Other): Extracorporeal Shock Wave Therapy to relieve pain after arthroscopy for osteochondral lesions of talus
  Interventions: Other: Extracorporeal Shock Wave Therapy

INTERVENTIONS:
Other: Extracorporeal Shock Wave Therapy — Extracorporeal Shock Wave Therapy will be used for pain-relief after arthroscopy for osteochondral lesions of the talus

SUMMARY:
Arthroscopic surgery is effective in treating osteochondral lesions of the talus. However, there are still some patients with postoperative ankle pain. This study aims to investigate the clinical efficacy of shock wave adjuvant therapy in the treatment of postoperative pain caused by cartilage injury of talus after arthroscopy and to provide basis for further popularization and application.

DETAILED DESCRIPTION:
Arthroscopic surgery is effective in treating osteochondral lesions of the talus. However, there are still some patients with postoperative ankle pain. This study was conducted to investigate the clinical efficacy of shock wave therapy in the treatment of postoperative pain caused by cartilage injury of talus after arthroscopy.

Patients with osteochondral lesions of the talus treated by arthroscopic microfracture surgery and still complained ankle pain three months after surgery were enrolled. Radial extracorporeal shock wave therapy was used to give energy to the injured region of the talus and the adjacent area.Treatment was done once a week for 5 consecutive weeks. After shock wave therapy,the patients were followed by Visual Analogue Scale (VAS), the American Orthopaedic Foot and Ankle Society ankle-hindfoot scale(AOFAS-AHFS) , and followed finally by Magnetic Resonance Imaging(MRI) of the ankle.

ELIGIBILITY:
Inclusion Criteria:

1. For arthroscopy:

   * Ankle pain, aggravated after exercise or weight-bearing activity, accompanied by lameness, joint stiffness and dysfunction for at least 3 months
   * No talar collapse
   * Talar cartilage injury cases before stage Ⅳ of Hepple classification
2. For shock wave therapy:

   * Patients with micro-fractures treated with arthroscopic treatment of talar cartilage injury and were treated with routine rehabilitation training after arthroscopy
   * Patients who till complained obvious ankle pain 3 months after surgery

Exclusion Criteria:

* Severe cardiovascular and cerebrovascular diseases
* Hemorrhagic diseases, coagulation disorders
* Bone immaturity
* Thrombosis
* Use of anti-immune agents
* Various types of tumor patients
* Pregnant women
* History of mental illness
* Patients who could not be followed
* Patients with other lower extremity injuries after surgery and were unwilling to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Change of VAS scores before and after shock wave therapy | 6 weeks, 12 weeks and last follow-up at an average of 2 years after shock wave therapy
  The Visual Analogue Scale scores of the patients before and after the shock wave therapy are recorded. The scale ranges from 0-10 points, and decreases of the value represent a better outcome. The data analyses are performed with SPSS version 16.0 statistical software. Continuous variables are expressed as mean ± standard deviation, and 95% confidence intervals are determined. The data are compared by paired t test or rank-sum test. P value < 0.05 is considered as statistically significant.

SECONDARY OUTCOMES:
Change of AOFAS scores before and after shock wave therapy | 6 weeks, 12 weeks and last follow-up last follow-up at an average of 2 years after shock wave therapy
  The American Orthopaedic Foot & Ankle Society scores of the patients before and after the shock wave therapy are recorded. The scale ranges from 0-100 points, and increases of the value represent a better outcome. The data analyses are performed with SPSS version 16.0 statistical software. Continuous variables are expressed as mean ± standard deviation, and 95% confidence intervals are determined. The data are compared by paired t test or rank-sum test. P value < 0.05 is considered as statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Duan, M.D., Principal Investigator — Southwest Hospital, China
Locations (1):
- Southwest Hospital, Chongqing, China

IPD SHARING:
Plan to Share IPD: No